CLINICAL TRIAL: NCT01666171
Title: Change in Mammographic Density With Metformin Use: A Companion Study to NCIC Study MA.32
Brief Title: Studying Changes in Breast Density in Patients With Early-Stage Breast Cancer Treated With Metformin Hydrochloride or Placebo on CAN-NCIC-MA.32
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cancer and Leukemia Group B (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Richard L. Schilsky, Cancer and Leukemia Group B
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CALGB-A211201; CDR0000738328 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: estrogen receptor-negative breast cancer; progesterone receptor-negative breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin; Watchful Waiting

INTERVENTIONS:
Drug: metformin hydrochloride
Other: clinical observation
Other: diagnostic laboratory biomarker analysis
Other: imaging biomarker analysis
Other: medical chart review
Procedure: digital mammography

SUMMARY:
RATIONALE: Learning about the effect of metformin hydrochloride in breast density of women with early-stage breast cancer may help plan treatment.

PURPOSE: This trial studies changes in breast density in patients with early-stage breast cancer treated with metformin hydrochloride or placebo on CAN-NCIC-MA.32.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the change in percent mammographic density in contralateral (unaffected breast) from prior to the initiation of metformin hydrochloride (metformin) or placebo treatment through one year of therapy in patients with hormone receptor-negative breast cancer (i.e., not on endocrine therapy).

Secondary

* To evaluate the change in percent breast density in contralateral (unaffected breast) from prior to the initiation of metformin or placebo treatment through two years of therapy in patients with hormone receptor-negative breast cancer (i.e., not on endocrine therapy).
* To evaluate whether baseline mammographic density correlates with baseline of fasting plasma insulin, glucose levels, and Homeostasis Model Assessment (HOMA) (collected on the treatment protocol CAN-NCIC-MA.32) (MA.32).
* To evaluate whether changes in dense area in response to metformin therapy from pre-treatment through two years of therapy correlate with changes in fasting plasma insulin, glucose levels, and HOMA (collected on the treatment protocol MA.32) over the same time period.
* To explore whether change in mammographic density for women on metformin is associated with risk of second primary breast cancer.

OUTLINE: Patients' mammograms taken at baseline and at approximately 1 and 2 years of metformin or placebo treatment are retrieved and analyzed for breast-density change. Pre-menopausal patients' menstrual cycle information is also collected at baseline and every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must either be concurrently enrolling or previously enrolled to Canada (CAN) National Cancer Institute of Canada (NCIC) study MA.32 (CAN-NCIC-MA.32) (MA.32); eligible patients may be either pre- or post-menopausal
* Patients must have hormone receptor-negative breast cancer
* Patients must have breast density ≥ 25% (correlating with the Breast Imaging-Reporting and Data [BIRAD]-2 category of "scattered fibroglandular densities" or greater)
* Baseline digital mammograms taken within 12 months prior to registration to MA.32, with at least a craniocaudal (CC) view used for enrollment to MA.32 must be available for submission; if the patient has previously enrolled to MA.32 and one year has elapsed from baseline mammograms, one-year mammograms must also be available for submission
* Contralateral unaffected breast in place (with no prior cancer or radiation, no implants, and no plan for breast surgery on contralateral breast over the course of the study); women with a prior biopsy on the unaffected breast are eligible

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Women receiving endocrine therapy (e.g., tamoxifen, aromatase inhibitors) are not eligible

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change in percent mammographic breast density in contralateral (unaffected) breast from baseline to 1 year using two-sample t-test or Wilcoxon rank-sum test

SECONDARY OUTCOMES:
Change in percent mammographic breast density in contralateral (unaffected) breast from baseline to 2 years using two-sample t-test
Correlation between baseline mammographic density and baseline plasma fasting insulin, glucose levels, and HOMA using a scatter plot, correlation-coefficient estimation, and linear-regression method
Correlation of changes in dense area in response to metformin therapy from pre-treatment to on treatment (at year 1 and year 2) with plasma fasting insulin, glucose levels, and HOMA using simple linear-regression method
Correlation between mammographic density and the incidence of second primary breast cancer using correlation coefficient and scatter plot

CONTACTS AND LOCATIONS:
Overall Officials: Marie E. Wood, MD, Principal Investigator — University of Vermont